CLINICAL TRIAL: NCT05689294
Title: Piezoelectric Sensors for Non-invasive Continuous Arterial Blood Pressure Measurements
Brief Title: Non Invasive Continuous Blood Pressure Sensor
Status: Completed | Type: Observational
Sponsor: Dartmouth-Hitchcock Medical Center (Other)
Collaborators: Dartmouth College (Other)
Responsible Party: Principal Investigator, Alexander T. Abess, Assistant Professor of Anesthesiology, Geisel School of Medicine, Dartmouth, Dartmouth-Hitchcock Medical Center
Other Study IDs: STUDY02001549
Record Dates: First submitted 2023-01-03; First posted 2023-01-19 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Blood Pressure; Arterial Line; Anesthesia
Keywords: Piezoelectric; Array Sensor; Blood Pressure; Monitoring; Arterial Line; Non-invasive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The primary objective of this study is to collect training data in order to establish a method for correlating arterial blood pressure with voltage output signals from a non-invasive piezoelectric array sensor placed on the skin superficial to the radial artery.

DETAILED DESCRIPTION:
The primary objective of this study is to collect training data in order to establish a method for correlating arterial blood pressure with voltage output signals from a non-invasive piezoelectric array sensor placed on the skin superficial to the radial artery. The development of this sensor could allow for non-invasive continuous measurement of arterial blood pressure.

The key hypothesis is: if the piezoelectric array sensor can detect pulsatile pressure waves when placed on a near surface artery and pulse wave analysis has been shown to allow for accurate beat-to-beat estimation of blood pressure, then the device placed superficial to a near surface artery should allow for the non-invasive estimation of continuous blood pressure.

Secondary objectives include identification of any significant ergonomic and motion artifact issues that could affect sensor utilization in future applications.

ELIGIBILITY:
Inclusion Criteria:

* Adults (18yr and older)
* Undergoing a planned (non-emergent, non-urgent) surgical procedure at DHMC for which an invasive arterial pressure monitor is standard clinical practice. Typical surgical procedures include but are not limited to craniotomy, thoracic surgery, abdominal surgery, and others.

Exclusion Criteria:

* Morbid obesity (BMI >40)
* Radial artery depth > 1cm from skin at location of sensor
* Peripheral vascular disease
* Atrial fibrillation
* Sensitivity or allergy to silicone or medical adhesive tape
* Inability to consent.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients undergoing elective surgery with planned utilization of invasive arterial pressure monitoring.
Sampling Method: Non-Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2023-04-01 (Actual); Primary Completion 2023-10-30 (Actual); Study Completion 2023-10-30 (Actual)

PRIMARY OUTCOMES:
Arterial Blood Pressure Measurement from Arterial Line | Surgery start to surgery stop
  We will be capturing arterial blood pressure measurement per standard of care from arterial line. This will include systolic and diastolic measurements and will be sampled continuously from standard invasive monitoring equipment. Because of the high frequency sampling, we will be capturing the entire pulse waveform with each heartbeat.
Arterial Blood Pressure Measurement from Non Invasive Sensor | Surgery start to surgery stop
  The piezoelectric sensor array detects mechanical pressure from the radial artery that is transmitted to the skin and converts this to microvolt electric potentials. These microvolt signals are captured by the sensor array equipment. The microvolt signals will be time-synchronized with the standard of care invasive arterial line pressure data.

SECONDARY OUTCOMES:
Assessment of accuracy of algorithm to convert piezoelectric signal data into blood pressure measurements. | Approximately 4 months following collection of data from subjects
  Approximately 80% of the data collected in this study will be used to refine and train an algorithm which has previously been validated on phantom and swine models to convert piezoelectric sensor data into meaningful blood pressure measurements. The remaining data (approximately 20%) will be used to test the accuracy of the algorithm against actual measured invasive blood pressure. Accuracy will be measured in terms of +/- mmHg at diastolic and systolic pressures.

CONTACTS AND LOCATIONS:
Overall Officials: Alexander T Abess, MD, Principal Investigator — Dartmouth-Hitchcock Medical Center
Locations (1):
- Dartmouth Hitchcock Medical Center, Lebanon, New Hampshire, United States

IPD SHARING:
Plan to Share IPD: No